CLINICAL TRIAL: NCT01826318
Title: Impact of a Stress Coping Strategy on Perceived Stress Levels and Performance During a Simulated Cardiopulmonary Resuscitation: A Randomized Controlled Trial
Brief Title: Stress Coping Strategy on Perceived Stress Levels and Performance During a Simulated Cardiopulmonary Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: SH_SIP_2007
Record Dates: First submitted 2013-04-03; First posted 2013-04-08 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Cardiopulmonary Resuscitations
Keywords: Stress; coping; simulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): Participants received a 10 minute instruction to cope with stress by loudly posing two task-focusing questions ("what is the patient's condition?", "what immediate action is needed?") when feeling overwhelmed by stress (intervention group)
  Interventions: Behavioral: Stress coping
- Control (No Intervention): Students in the control group did not receive any further instructions.

INTERVENTIONS:
Behavioral: Stress coping — Students in the intervention group received a 10 minute instruction to cope with stress. They were informed that an emergency situation is a stressful experience for health care workers and that perceived stress may interfere with their decision-making abilities and performance. Particularly, feeling overwhelmed by stress may cause cognitive impairment potentially leading to loss of concept how to deal with an emergency situation, which in turn further increases stress (vicious cycle). However, it is possible to overcome this situation by focusing on the basic conditions of the situation and the immediate actions that are needed. They were instructed that they should ask two task-focusing questions aloud ("what is the patient's condition?", "what immediate action is needed?") to overcome the negative consequences of feeling overwhelmed by stress.
  Arms: intervention

SUMMARY:
This study assessed the impact of a task-focusing strategy on perceived stress levels and performance during a simulated CPR scenario.

DETAILED DESCRIPTION:
Background: Cardiopulmonary resuscitation (CPR) causes significant stress, which may cause deficiencies in attention and increase distractibility. This may lead to misjudgements of priorities and delays in CPR performance, which may further increase mental stress (vicious cycle).

Aim: This study assessed the impact of a task-focusing strategy on perceived stress levels and performance during a simulated CPR scenario.

Methods: This is a prospective, randomized-controlled trial

Setting: Simulator-center of the University Hospital Basel, Switzerland.

Participants: A total of 124 volunteer medical students

Intervention: Randomization to receive a 10 minute instruction to cope with stress by loudly posing two task-focusing questions ("what is the patient's condition?", "what immediate action is needed?") when feeling overwhelmed by stress (intervention group) or a control group.

Outcome measures: The primary outcome is the perceived levels of stress and feeling overwhelmed (stress/overload); secondary outcomes were hands-on time, time to start CPR and number of leadership statements.

ELIGIBILITY:
Inclusion Criteria:

* 4th year medical students

Exclusion Criteria:

* none

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2007-12; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Average level of stress/overload during the resuscitation period | In the first 120 seconds after the onset of the cardiac arrest
  The primary outcome was the average level of stress/overload during the resuscitation period for the experimental and the control group.

SECONDARY OUTCOMES:
hands-on time | in the first 120 seconds after the onset of the cardiac arrest.
  Medical performance measures: hands-on time defined as duration of uninterrupted chest compressions and defibrillation in the first 120 seconds after the onset of the cardiac arrest.
time elapsed until CPR was started | in the first 120 seconds after the onset of the cardiac arrest
  the time elapsed until CPR was started, defined as the time to the first meaningful measure (either defibrillation, chest compression or ventilation) after the onset of the cardiac arrest; the team coordination measure
leadership statements | in the first 120 seconds after the onset of the cardiac arrest
  Number of leadership statements coded, using a predefined checklist containing the following categories based on previous research

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Hunziker, MD, MPH, Principal Investigator — University Hospital Basel, Basel 4031 Basel, Switzerland
Locations (1):
- University Hospital Basel, ICU, Basel, Canton of Basel-City, Switzerland